CLINICAL TRIAL: NCT04616729
Title: DEPO-Trigger Trial: GnRH Agonist DEPOt TRIGGER for Final Oocyte Maturation in Breast Cancer Patients Undergoing Fertility Preservation: a Pilot Study
Brief Title: DEPO-Trigger Trial: GnRH Agonist DEPOt TRIGGER for Final Oocyte Maturation
Acronym: Depo-Trigger
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universitair Ziekenhuis Brussel (Other)
Collaborators: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2019DEPO-TRIGGER001
Record Dates: First submitted 2020-10-21; First posted 2020-11-05 (Actual); Last update posted 2023-05-18 (Actual); Status verified 2023-04

CONDITIONS: Breast Cancer Female
Keywords: Fertility preservation; Reproductive Techniques, assisted; Ovulation Induction; Oocyte Retrieval; Cryopreservation
MeSH Terms: conditions — Helping Behavior | interventions — Triptorelin Pamoate; Injections

STUDY DESIGN:
Intervention Model Description: Patients will be randomized before start of ovarian stimulation to either DEPOT group (group A) or control group (group B), only after patient eligibility has been established and patient consent has been obtained.
  Group A will receive the GnRH agonist Depot form for final oocyte maturation followed by daily GnRH antagonist injections for 1 week.
  Group B will receive the GnRH agonist daily form for final oocyte maturation. After one week the Depot form combined with daily GnRH antagonist injections for 7 days, will be administered in view of ovarian protection during chemotherapy.
  Blood analysis and ultrasounds will be organised on day 3, 5 and 7 after oocyte pick-up in both groups.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- GnRH agonist Depot form (Experimental): Ovarian stimulation will be performed using a fixed antagonist protocol with Follitropin Alfa (daily in the evening) and Ganirelix or Cetrorelix (daily in the morning). Selection of the daily gonadotropin dose will be based on ovarian reserve parameters (AMH and AFC) and BMI. Co-administration of 5 mg of letrozole daily (in the morning) commencing on the first day of gonadotropin administration and continuing throughout the ovarian stimulation will be performed as this reduces oestradiol concentrations. GnRH agonist Triptorelin 3.75 mg Depot form will be used for final oocyte maturation. Ganirelix/Cetrorelix 0.25mg daily (in the morning) will resume for 7 days from the evening of the day of oocyte retrieval onwards. Hormone analysis, analysis of haematology and biochemistry and a pelvic ultrasound scan will be done on days 3, 5 and 7 after oocyte retrieval.
  Interventions: Drug: Triptorelin 3.75 MG Injection; Procedure: Transvaginal oocyte retrieval
- GnRH agonist Daily form (Active Comparator): Ovarian stimulation will be performed using a fixed antagonist protocol with Follitropin Alfa (daily in the evening) and Ganirelix/Cetrorelix (daily in the morning). Selection of the daily gonadotropin dose will be based on ovarian reserve parameters (AMH and AFC) and BMI. Co-administration of 5 mg of letrozole daily (in the morning) commencing on the first day of gonadotropin administration and continuing throughout the ovarian stimulation will be performed as this reduces oestradiol concentrations. GnRH agonist Triptorelin 0.2 mg Daily form will be used for final oocyte maturation. Hormone analysis, analysis of haematology and biochemistry and a pelvic ultrasound scan will be done on days 3, 5 and 7 after oocyte retrieval. The first administration of Triptorelin 3.75mg depot will be scheduled on the first day of the menstrual cycle after oocyte retrieval. To prevent the flare-up produced by the GnRH agonist, daily doses of 0.25mg of Ganirelix/Cetrorelix will be given for seven days.
  Interventions: Procedure: Transvaginal oocyte retrieval; Drug: Triptorelin Injection

INTERVENTIONS:
Drug: Triptorelin 3.75 MG Injection — Depot Group (Group A) will receive Triptorelin 3.75mg Depot form for final oocyte maturation.
  Other Names: Gonapeptyl; Decapeptyl
  Arms: GnRH agonist Depot form
Procedure: Transvaginal oocyte retrieval — Patients in both groups will undergo a transvaginal oocyte retrieval after ovarian stimulation.
Drug: Triptorelin Injection — Daily Group (Group B) will receive Triptorelin 0.2mg Daily form for final oocyte maturation.
  Other Names: Gonapeptyl; Decapeptyl
  Arms: GnRH agonist Daily form

SUMMARY:
For breast cancer patients who are candidates to receive chemotherapy, concurrent use of temporary ovarian suppression with gonadotropin-releasing hormone agonists (GnRHa) can be offered as ovarian protection.

Because ovarian stimulation for oocyte cryopreservation is usually performed using a GnRH antagonist protocol and typically involves final oocyte maturation triggering with a GnRH agonist, the investigators designed this study to explore the feasibility of combining the final oocyte maturation trigger and the start of ovarian suppression. Short-term cotreatment with GnRH antagonists is needed to induce rapid luteolysis (in view of prevention of ovarian hyperstimulation).

To demonstrate the safety of GnRH agonist depot triggering followed by daily GnRH antagonist luteolysis, this pilot study is set out to analyse the endocrine profile and ovarian morphology of this novel protocol.

DETAILED DESCRIPTION:
For breast cancer patients who are candidates to receive chemotherapy, concurrent use of temporary ovarian suppression with gonadotropin-releasing hormone agonists (GnRHa) can be offered as ovarian protection. A recent meta-analysis of individual patient data from the largest randomised clinical trials in women with early breast cancer indicated beneficial effects of GnRHa ovarian suppression in reducing POI risk and increasing post-chemotherapy pregnancy rates with no negative effect on patients' outcomes. However, it should not be considered as an alternative to cryopreservation strategies in fertility preservation.

Because ovarian stimulation for oocyte cryopreservation is usually performed using a GnRH antagonist protocol and typically involves final oocyte maturation triggering with a GnRH agonist, the investigators designed this study to explore the feasibility of combining the final oocyte maturation trigger and the start of ovarian suppression. Replacement of the 0,2mg triptorelin trigger by a GnRH agonist depot has potential to provide this dual action. However, the protracted action of the GnRH agonist depot will result in prolonged stimulation of multiple corpora lutea, which will lead to enhanced production of steroids (estradiol and progesterone) and growth factors such as vascular endothelial growth factor. Consequently, GnRH agonist-induced stimulation of multiple corpora lutea is potentially unsafe in a patient with breast cancer because of the impact of estradiol and progesterone on breast tumour cells. In addition, VEGF may increase the risk of OHSS, which will lead to postponement of cancer treatment. Therefore, short-term cotreatment with GnRH antagonists is needed to induce rapid luteolysis.

To demonstrate the safety of GnRH agonist depot triggering followed by daily GnRH antagonist luteolysis, this pilot study is set out to analyse the endocrine profile and ovarian morphology of this novel protocol.

Patients will be randomized before start of stimulation to either DEPOT group (group A) or control group (group B), only after patient eligibility has been established and patient consent has been obtained.

ELIGIBILITY:
Inclusion Criteria:

* Age <36y
* BMI ≥ 18 and ≤ 35 kg/m²
* Early stage breast cancer
* Any hormone receptor status
* Any HER status
* Cryopreservation of oocytes and/or embryos
* Oncologist's approval to participate to the DEPO-trigger trial
* Signed informed consent form

Exclusion Criteria:

* Contra-indications for controlled ovarian stimulation or oocyte retrieval
* Necessity of neo-adjuvant chemotherapy

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2022-11-01 (Actual); Primary Completion 2025-11-30 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Safety profile with regard to the risk of OHSS: assessment of change in ovarian volume | During one week after the transvaginal oocyte retrieval (on day 3, 5 and 7)
  A transvaginal ultrasound will be performed to measure the ovarian volume according to the formula 'length x width x height x 0.523' mm³.
  In the assumption of safety ovarian volume should be similar to that in the control group and there should be no events of ovarian hyperstimulation syndrome.
Safety profile with regard to the risk of OHSS: assessment of change in hematocrit | During one week after the transvaginal oocyte retrieval (on day 3, 5 and 7)
  A blood sample will be taken to evaluate hematocrit (%). In the assumption of safety hematocrit levels should be similar to that in the control group and there should be no events of ovarian hyperstimulation syndrome.
Safety profile with regard to the risk of OHSS: assessment of change in hemoglobine | During one week after the transvaginal oocyte retrieval (on day 3, 5 and 7)
  A blood sample will be taken to evaluate hemoglobine (g/dL). In the assumption of safety hemoglobine levels should be similar to that in the control group and there should be no events of ovarian hyperstimulation syndrome.
Safety profile with regard to the risk of OHSS: assessment of change in White Blood cell Count | During one week after the transvaginal oocyte retrieval (on day 3, 5 and 7)
  A blood sample will be taken to evaluate White Blood cell Count (X10³/mm³). In the assumption of safety White Blood cell Count should be similar to that in the control group and there should be no events of ovarian hyperstimulation syndrome.
Safety profile with regard to the risk of OHSS: assessment of change in Platelet Count | During one week after the transvaginal oocyte retrieval (on day 3, 5 and 7)
  A blood sample will be taken to evaluate Platelet Count (X10³/mm³). In the assumption of safety Platelet Count should be similar to that in the control group and there should be no events of ovarian hyperstimulation syndrome.
Safety profile with regard to the risk of OHSS: assessment of change in estimated glomerular filtration rate (eGFR) | During one week after the transvaginal oocyte retrieval (on day 3, 5 and 7)
  A blood sample will be taken to evaluate eGFR (mL/min/1.73m²). In the assumption of safety eGFR levels should be similar to that in the control group and there should be no events of ovarian hyperstimulation syndrome.
Safety profile with regard to the risk of OHSS: assessment of change in Creatinine | During one week after the transvaginal oocyte retrieval (on day 3, 5 and 7)
  A blood sample will be taken to evaluate Creatinine (mg/dL). In the assumption of safety creatinine levels should be similar to that in the control group and there should be no events of ovarian hyperstimulation syndrome.
Safety profile with regard to the risk of OHSS: assessment of change in Albumin | During one week after the transvaginal oocyte retrieval (on day 3, 5 and 7)
  A blood sample will be taken to evaluate Albumin (g/L). In the assumption of safety Albumin levels should be similar to that in the control group and there should be no events of ovarian hyperstimulation syndrome.
Safety profile with regard to the risk of OHSS: assessment of change in liver function (AST, ALT, Gamma-GT, bilirubine, LDH) | During one week after the transvaginal oocyte retrieval (on day 3, 5 and 7)
  A blood sample will be taken to evaluate liver function (AST U/L, ALT U/L, Gamma-GT U/L, bilirubine mg/dL, LDH U/L).
  In the assumption of safety liver function levels should be similar to that in the control group and there should be no events of ovarian hyperstimulation syndrome.
Safety profile with regard to the risk of OHSS: assessment of change in Oestradiol (E2) | During one week after the transvaginal oocyte retrieval (on day 3, 5 and 7)
  A blood sample will be taken to evaluate Oestradiol (ng/L). In the assumption of safety Oestradiol levels should be similar to that in the control group and there should be no events of ovarian hyperstimulation syndrome.
Safety profile with regard to the risk of OHSS: assessment of change in Progesteron | During one week after the transvaginal oocyte retrieval (on day 3, 5 and 7)
  A blood sample will be taken to evaluate Progesteron (mcg/L). In the assumption of safety Progesteron levels should be similar to that in the control group and there should be no events of ovarian hyperstimulation syndrome.
Safety profile with regard to the risk of OHSS: assessment of change in Follicle Stimulating Hormone (FSH) | During one week after the transvaginal oocyte retrieval (on day 3, 5 and 7)
  A blood sample will be taken to evaluate FSH (IU/L). In the assumption of safety FSH levels should be similar to that in the control group and there should be no events of ovarian hyperstimulation syndrome.
Safety profile with regard to the risk of OHSS: assessment of change in Luteinizing Hormone (LH) | During one week after the transvaginal oocyte retrieval (on day 3, 5 and 7)
  A blood sample will be taken to evaluate LH (IU/L). In the assumption of safety LH levels should be similar to that in the control group and there should be no events of ovarian hyperstimulation syndrome.

SECONDARY OUTCOMES:
Number of cumulus-oocyte complexes | During the procedure of the transvaginal oocyte retrieval
  Evaluation of the number of cumulus-oocyte complexes between the Depot Group and Daily Group
Number of Metaphase II oocytes | Immediately after the procedure of the transvaginal oocyte retrieval
  Evaluation of the number of Metaphase II oocytes between the Depot group and Daily group
Evaluation of climacteric symptoms | One week after the transvaginal oocyte retrieval (on day 7)
  Assessment of MENQOL (The Menopause-Specific Quality of Life) Questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Michel De Vos, MD PhD, Principal Investigator — Universitair Ziekenhuis Brussel
Locations (2):
- Belgium (2):
  - Universitair Ziekenhuis Brussel, Boortmeerbeek, Brussels Capital
  - Universitaire Ziekenhuizen Leuven, Leuven, Vlaams-Brabant

IPD SHARING:
Plan to Share IPD: Yes
As this is a multicenter study, we plan to share IPD between the study sites. An electronically case report form (eCRF) will be set up and completed in all sites. Data will be handled in accordance with the general data protection regulation (GDPR).
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: The data will become available over the course of the study until 6 months after ending this study. This will give us the time to analyse the data of the different sites.
Access Criteria: eCRF

REFERENCES:
- [Background] Lambertini M, Cinquini M, Moschetti I, Peccatori FA, Anserini P, Valenzano Menada M, Tomirotti M, Del Mastro L. Temporary ovarian suppression during chemotherapy to preserve ovarian function and fertility in breast cancer patients: A GRADE approach for evidence evaluation and recommendations by the Italian Association of Medical Oncology. Eur J Cancer. 2017 Jan;71:25-33. doi: 10.1016/j.ejca.2016.10.034. Epub 2016 Dec 9. PMID 27940355
- [Background] Lambertini M, Moore HCF, Leonard RCF, Loibl S, Munster P, Bruzzone M, Boni L, Unger JM, Anderson RA, Mehta K, Minton S, Poggio F, Albain KS, Adamson DJA, Gerber B, Cripps A, Bertelli G, Seiler S, Ceppi M, Partridge AH, Del Mastro L. Gonadotropin-Releasing Hormone Agonists During Chemotherapy for Preservation of Ovarian Function and Fertility in Premenopausal Patients With Early Breast Cancer: A Systematic Review and Meta-Analysis of Individual Patient-Level Data. J Clin Oncol. 2018 Jul 1;36(19):1981-1990. doi: 10.1200/JCO.2018.78.0858. Epub 2018 May 2. PMID 29718793